CLINICAL TRIAL: NCT05805995
Title: Impact of Vertebral Derotation on Ventilatory Functions and Chest Circumference in Adolescent Scoliosis
Brief Title: Effects of Vertebral Derotation on Pulmonary Functions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Khaled Takey Ahmed, Asssociate Professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: veretebral derotation
Record Dates: First submitted 2023-03-28; First posted 2023-04-10 (Actual); Last update posted 2023-04-10 (Actual); Status verified 2023-03

CONDITIONS: Adolescent Idiopathic Scoliosis; Scoliosis Idiopathic
Keywords: lung functions, vertebral derotation, chest intervention

STUDY DESIGN:
Intervention Model Description: The exercise group received vertebral derotation with posterior correction in addition to routine chest physiotherapy (group A).
  The Control group received only posterior correction with routine chest physiotherapy (group B).
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- intervention group (Experimental): The exercise group received vertebral derotation with posterior correction in addition to routine chest physiotherapy (group A).
  Interventions: Procedure: vertebral derotation
- control (Experimental): The Control group received only posterior correction with routine chest physiotherapy (group B).
  Interventions: Procedure: vertebral derotation

INTERVENTIONS:
Procedure: vertebral derotation — * Incentive spirometer (Mediciser): Used for breathing exercises.
  * Cycle ergometer ( Mijnhardt , St. Paul, MN): Used for lower limb exercise.
  Other Names: INCENTIVE SPIROMETER

SUMMARY:
This study was conducted to determine the physiological and mechanical effects of physical training post surgical correction of adolescent scoliosis using vertebral derotation.

DETAILED DESCRIPTION:
Sixty patients from both sexes with idiopathic scoliosis underwent posterior correction (fusion). They were presented with idiopathic scoliosis for 6-12 month. Their mean Cobb's angle was measured in degrees and their mean angle of rotation was measured also in degrees. Before participation all the patients were examined clinically by a chest physician to exclude any cardio pulmonary or vascular disorders which may alter the pulmonary functions. All of them did not receive any physical therapy program prior to the operation.

Patients were arranged randomly into two groups (1 and 2), each containing 30 patients. Group 1 (DRG) received posterior correction, vertebral derotation technique during posterior correction and pulmonary rehabilitation program while group 2 (NDRG) received posterior correction and the same rehabilitation program given to group 1.

ELIGIBILITY:
Inclusion Criteria:

* Male patients suffering from adolescent idiopathic scoliosis.
* Participant age ranged from 12- 18 years old.
* All patients had the same medical care.
* Participants have received a good explanation of the treatment and measurement device.
* Treatment was conducted surgical intervention.

Exclusion Criteria:

* Instability of patient's medical condition.
* Presence of any diseases that could affect the study results.
* Participants having respiratory, cardiac, or neurological diseases that affect pulmonary functions.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-05-30 (Estimated); Study Completion 2023-06-15 (Estimated)

PRIMARY OUTCOMES:
(FEV1 and MVV) were measured by using the spirometer Pulmonary functions testing | Five months
  Each patient's weight in kilograms, and height in meters were recorded and entered the machine. An individual sat in a chair and inhaled deeply before closing their mouth tightly around the tube. Several exercises were carried out until the patient comprehended and was comfortable with the instruction. The patient inhaled deeply and exhaled as quickly as possible into the spirometer(Morgan Trans Flow Test Vicatest p2 (Kent, ME 87 ED, England).

CONTACTS AND LOCATIONS:
Locations (2):
- Egypt (2):
  - Faculty of Physical Therapy -Cu, Giza
  - faculty of PT - cu, Giza

IPD SHARING:
Plan to Share IPD: Yes
At first study protocol and informed consent
Supporting Information: Study Protocol, SAP, ICF
Time Frame: January 2023 - June 2023
Access Criteria: consent

REFERENCES:
- [Background] Kim YJ, Lenke LG, Bridwell KH, Kim KL, Steger-May K. Pulmonary function in adolescent idiopathic scoliosis relative to the surgical procedure. J Bone Joint Surg Am. 2005 Jul;87(7):1534-41. doi: 10.2106/JBJS.C.00978. PMID 15995121